CLINICAL TRIAL: NCT07179705
Title: Hypotension Prediction Index Guided Prevention of Intradialytic Hypotension During Intermittent Renal Replacement Therapy in Intensive Care Units
Brief Title: Using a Hypotension Prediction Index to Prevent Low Blood Pressure During Dialysis in ICU Patients
Acronym: HyPIR-ICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 0204/68
Record Dates: First submitted 2025-07-21; First posted 2025-09-18 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Intradialytic Hypotension; Intensive Care Unit ICU; Hemodialysis Patients
Keywords: Hypotension Prediction Index (HPI); Prolonged intermittent renal replacement therapy (PIRRT); Slow-low efficiency dialysis; Intradialytic hypotension; Hemodynamic monitoring; Intensive Care Unit

STUDY DESIGN:
Intervention Model Description: Study Design
  * Crossover design: Each participant receives both interventions (HPI-guided and standard care) during two dialysis sessions, with a 1-2 day washout between sessions.
  * Randomization: Block randomization stratified by kidney status (AKI vs. ESKD) and vasopressor use.
  * Open-label: Clinicians and participants are aware of the treatment; however, data analysis is blinded and performed independently.
  Intervention Arm A: HPI-guided management during first PIRRT → standard care in second session Arm B: Standard care during first PIRRT → HPI-guided management in second session
Who Masked: Outcomes Assessor
Masking Description: Clinicians and participants are aware of the treatment; however, data analysis is blinded and performed independently.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPI first (Experimental): Arm A: HPI-guided management during first PIRRT → standard care in second session
  Interventions: Device: Hypotensive prediction index
- Standard of care first (Experimental): Arm B: Standard care during first PIRRT → HPI-guided management in second session
  Interventions: Device: Standard of care monitoring

INTERVENTIONS:
Device: Hypotensive prediction index — The HPI, developed by Edwards Lifesciences and integrated into the HemosphereⓇ hemodynamic monitoring system, is an algorithm-based tool that predicts hypotensive events before they occur, allowing earlier intervention. While this tool has shown benefit in surgical and post-operative settings, it has not been tested in ICU patients undergoing dialysis.
  Arms: HPI first
Device: Standard of care monitoring — Standard of Care
  * Monitoring via conventional invasive BP and clinical judgment
  * Use of physical exam, CVP, PPV, and response-based decisions (fluid bolus, vasopressors)
  Arms: Standard of care first

SUMMARY:
This single-center, crossover randomized controlled trial (HyPIR-ICU) investigates whether a Hypotension Prediction Index (HPI)-guided management strategy can reduce intradialytic hypotension (IDH) during prolonged intermittent renal replacement therapy (PIRRT) in critically ill patients. All participants must have an indwelling arterial catheter for continuous hemodynamic monitoring.

DETAILED DESCRIPTION:
This study explores whether HPI-guided management during PIRRT can randomization: Block randomization stratified by kidney status (AKI vs. ESKD) and vasopressor use. All parameters are monitored in real-time via the HemosphereⓇ system and reassessed after each intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years old
* Diagnosed with acute kidney injury (AKI) or end-stage kidney disease (ESKD)
* Admitted to medical ICU
* Scheduled for PIRRT
* Have an indwelling arterial catheter

Exclusion Criteria:

* Severe right heart dysfunction, significant valvular disease, arrhythmias, mechanical circulatory support, absence of arterial access, no UF prescription, palliative care, or expected ICU stay <72 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
- Time-weighted average mean arterial pressure <65 mmHg (TWA-MAP<65 mmHg) | Day 1 and Day 3
  Average intensity and duration of time that a patient's mean arterial pressure (MAP) falls below 65 mmHg, which is considered the critical threshold for maintaining adequate organ perfusion.

SECONDARY OUTCOMES:
Intradialytic hypotension frequency by various definitions | Day 1 and Day 3
  * Nadir90: Minimal intra-hemodialytic SBP<90 mmHg
  * Fall20: Pre-hemodialysis SBP - Minimal intra-hemodialytic SBP >20 mmHg
  * Fall20Nadir90: Meet criteria for Nadir 90 and Fall20
  * HEMO: Fall in SBP resulting in intervention of UF reduction, blood flow reduction, or intervention administration
Delivered UF/Prescribed UF | Day 1 and Day 3
  * Prescribed UF (Ultrafiltration): The amount of fluid (in milliliters or liters)
  * Delivered UF: The actual amount of fluid successfully removed during the session.
  * This ratio reflects the efficacy of fluid removal.
Incidence of tachycardia or significant arrhythmia | Day 1and Day 3
  Incidence of tachycardia or significant arrhythmia: defined by HR>130 bpm or HR increase >20% from pre-hemodialysis baseline for >15 min
Reaction time to treatment | Day 1 and Day 3
  Reaction time to treatment refers to the interval between the detection of a hypotensive event (or risk of it) and the initiation of appropriate clinical intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Nephrology, Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No